CLINICAL TRIAL: NCT03760406
Title: Optimization of VIM Targeting in Essential Tremor Surgery
Acronym: Opti-VIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CHUBX 2018/32
Record Dates: First submitted 2018-11-26; First posted 2018-11-30 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Essential Tremor
Keywords: Essential Tremor; Deep brain stimulation; Ventro-intermediate nucleus of the thalamus; Targeting; Asleep surgery
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Severe essential tremor treated by DBS (Experimental)
  Interventions: Procedure: Opti-VIM targeting in DBS surgery

INTERVENTIONS:
Procedure: Opti-VIM targeting in DBS surgery — DBS surgery will be performed under general anaesthesia, without intra-operative clinical and electrophysiological testing, with a surgical robot and under CT-scan guidance (O-Arm ©). The VIM coordinates will be calculated with the probabilistic model that have been developed.

SUMMARY:
Deep brain stimulation (DBS) for essential tremor is based on the intermedius ventralis nucleus of the thalamus (VIM) stimulation. This structure is however very difficult to target, as it remains invisible on imaging. The current procedure based on awake surgery with clinical and electrophysiological testings has several limitations that lead us to develop a probabilistic model to locate precisely the target. This study aims to show that asleep DBS surgery based on this new targeting method leads to at least the same clinical results than the classical procedure.

DETAILED DESCRIPTION:
The intermedius ventralis nucleus of the thalamus (VIM), which represents the target for deep brain stimulation (DBS) in essential tremor, still remains invisible on 1,5 tesla MRI (the only magnetic field available for stereotactic surgery). The target coordinates currently used are based on stereotactic atlases or mean coordinates from retrospective series. They are so imprecise that intra-operative clinical testing and micro-electrode recordings are mandatory to locate the exact position of the VIM. This procedure is long lasting, requires that the patient is awake, and increases the risk of intracerebral haemorrhage and nosocomial infections. Furthermore, some patients are not improved despite a DBS lead implanted in the electrophysiologically and clinically defined target. To overcome these limitations, investigators developed a probabilistic model based on data extracted from imaging of patients with particularly good outcomes after DBS surgery. This machine-learning model allows calculating to coordinates of the VIM according to the position of radio-anatomical landmarks with a mean precision of 1,65mm.

The aim of this study is to validate this new targeting method on a prospective cohort of patients. DBS surgery will be performed under general anaesthesia, without intra-operative clinical and electrophysiological testing, with a surgical robot and under CT-scan guidance (O-Arm ©).

Neurostimulation device programming will be performed as usual. Patients' tremor and quality of life will be evaluated pre and post-operatively at 3 months, according to the Fahn-Tolosa-Marin (FTM) scale and with an accelerometry recording (for tremor) and with the mPDQ-39 scale for quality of life. Surgical complications and side effects related to neurostimulation will be gathered all along the follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Severe essential tremor despite the optimal medical management
* Age between 18 and 75 years
* Normal MRI scan
* Mattis Dementia Rating Scale (MDRS) score ≥ 130
* Affiliation to the social security
* Signed informed consent

Exclusion Criteria:

* Depression (Beck Depression Inventory scale > 20)
* Contra-indication to surgery or general anesthesia
* Cerebral atrophy on MRI scan
* Pregnant or breastfeeding women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2023-08-29 (Actual); Study Completion 2023-08-29 (Actual)

PRIMARY OUTCOMES:
Change of Fahn-Tolosa-Marin (FTM) scale score | Before and 3 month after DBS surgery
  Scale global range : min=0 / max=160 Higher values represent worse tremor

SECONDARY OUTCOMES:
Accelerometry recordings : spectral analysis | Before and 3 month after DBS surgery
  Accelerometry recordings at the pre-inclusion visit and at 3 months after surgery in ON and OFF-stimulation conditions with spectral analysis.
Accelerometry recordings : calculation of the total accelerometry power | Before and 3 month after DBS surgery
  Accelerometry recordings at the pre-inclusion visit and at 3 months after surgery in ON and OFF-stimulation conditions with calculation of the total accelerometry power.
Surgical complications | Up to 3 month after DBS surgery
  Onset of infection, hematoma or seizure
Device complications and dysfunction | Up to 3 month after DBS surgery
  rupture or displacement of electrode, pain at the stimulation box implantation site or along the subcutaneous cable if they require further intervention, infection.
Neurostimulation-related side effects | Up to 3 month after DBS surgery
  Onset of dysarthria and ataxia assessed by the items 1 to 4 of the Scale for Assessment and Rating of Ataxia (SARA), ataxia assessed by a posturometry analysis, paresthesia, muscular contractions
Quality of life: change of modified Parkinson's Disease Questionnaire-39 (mPDQ-39) scale score | Before and 3 month after DBS surgery
  Adaptation of Parkinson's Disease Questionnaire-39 to essential tremor Scale global range : min=0 / max=156 Higher values represent worse Quality of life
Coordinates of active contacts | 3 month after DBS surgery
  Coordinates of active contacts (i.e; the contact with the best effect on tremor without side effects) These coordinates (x, y, z) are obtained by merging the images of the 3-month postoperative scanner with the images of the preoperative MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Antoine BENARD, MD, Study Chair — USMR CHU de Bordeaux
Locations (2):
- France (2):
  - CHU de Bordeaux, Bordeaux
  - Hospices Civils de Lyon, Bron